CLINICAL TRIAL: NCT06805942
Title: Embolization for the Treatment of Heel Pain Secondary to Plantar Fasciitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IR Centers (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12382
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Plantar Fasciitis of Both Feet
MeSH Terms: interventions — Injections

STUDY DESIGN:
Intervention Model Description: This study uses a single-group assignment model where all enrolled participants will receive the same intervention, plantar fascia embolization (PFE) with Lipiodol, to evaluate its safety, feasibility, and effectiveness for treating plantar fasciitis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single Intervention Group (Experimental): Participants in this arm will receive plantar fascia embolization (PFE) using Lipiodol (ethiodized oil) to treat pain caused by plantar fasciitis.
  Interventions: Device: Lipiodol (ethiodized oil) injection

INTERVENTIONS:
Device: Lipiodol (ethiodized oil) injection — Lipiodol will be used as an embolic agent for arterial embolization targeting neovascularity in the plantar fascia to reduce inflammation and pain.

SUMMARY:
This study evaluates the feasibility and safety of using Lipiodol (ethiodized oil) as an investigational embolic agent for treating pain caused by plantar fasciitis. Participants will undergo a minimally invasive procedure called plantar fascia embolization (PFE) to reduce inflammation and pain in the affected area. The study aims to assess changes in pain levels, foot function, and any potential side effects over a six-month follow-up period.

DETAILED DESCRIPTION:
This study investigates the use of Lipiodol (ethiodized oil) for plantar fascia embolization (PFE) to treat pain from plantar fasciitis. It focuses on evaluating safety, feasibility, and outcomes related to pain reduction and improved foot function.

ELIGIBILITY:
Inclusion Criteria:Participants aged 22 years or older. Diagnosed with plantar fasciitis by an orthopedic or podiatry surgeon.

Ultrasound evaluation showing:

Increased plantar fascia thickness > 4 mm. Hyperemia in the plantar fascia near its proximal insertion or perifascial soft tissue.

Self-reported pain of at least 5/10 on the Visual Analog Scale (VAS). Negative X-ray for acute fractures. Refractory to at least 6 weeks of conservative therapies. Able to provide written informed consent. -

Exclusion Criteria:Heel pain caused by stress fractures, nerve entrapment, or inflammatory conditions such as arthritis, gout, or bursitis.

Corticosteroid injection in the plantar fascia within 90 days prior to embolization.

Prior surgical repair or plantar fascia rupture. Severe allergy to Lipiodol or iodinated contrast media. Diagnosis of peripheral arterial disease affecting the lower extremities. Active workers' compensation claim for plantar fasciitis. Pregnancy or breastfeeding. Type 1 Diabetes Mellitus or significant renal dysfunction (GFR < 45 or serum creatinine > 2.0 mg/dL).

Sensory or motor neuropathy of the feet. Active skin wounds on the plantar surface of the affected foot.

-

Ages: 22 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in Pain (VAS Score) | Baseline to 6 months
  Change in pain level as measured by the Visual Analog Scale (VAS), with scores ranging from 0 (no pain) to 10 (worst pain imaginable).

SECONDARY OUTCOMES:
Improvement in Foot Function (FAAM Score) | Baseline to 6 months
  Change in function as assessed by the Foot and Ankle Ability Measure (FAAM), including activities of daily living and sports subscales.

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Bagla, MD, Principal Investigator — IR Centers
Locations (1):
- IR Centers, Falls Church, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gandhi R, Banker M. Early outcomes of transcatheter arterial embolization using imipenem/cilastatin for plantar fasciitis refractory to conservative therapy. Br J Radiol. 2024 Feb 28;97(1155):544-548. doi: 10.1093/bjr/tqae012. PMID 38281074
- [Result] Sasaki T, Shibuya M, Miyazaki K, Nakata M, Kawabe A, Nakasone T, Sakai N, Okuno Y. Clinical results of ultrasound-guided intra-arterial embolization targeting abnormal neovessels for plantar fasciitis: 66 cases with up to 4 years of follow-up. Foot Ankle Surg. 2025 Feb;31(2):105-110. doi: 10.1016/j.fas.2024.07.009. Epub 2024 Jul 27. PMID 39089905
- [Result] Sapoval M, Querub C, Pereira H, Pellerin O, Boeken T, Di Gaeta A, Ahmar MA, Lefevre-Colau MM, Nguyen C, Daste C, Lacroix M, Laredo JD, Sabatier B, Martelli N, Chatellier G, Dean C, Rannou F. Genicular artery embolization for knee osteoarthritis: Results of the LipioJoint-1 trial. Diagn Interv Imaging. 2024 Apr;105(4):144-150. doi: 10.1016/j.diii.2023.12.003. Epub 2023 Dec 14. PMID 38102013